CLINICAL TRIAL: NCT04783454
Title: Preventing Neck & Back Pain in Teleworking Office Workers: a Randomized Controlled Trial
Acronym: Prevent@HOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BC-08635
Record Dates: First submitted 2021-02-26; First posted 2021-03-05 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain; Low Back Pain; Back Pain
Keywords: desktop workers; telework; remote work; sedentary work; primary prevention
MeSH Terms: conditions — Neck Pain; Low Back Pain; Back Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: All investigators and outcome assessors are blind to the subjects' allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): * single (online) educational video on how the prevention program is designed and general advice on (how to adopt) a healthy lifestyle
  * 12-week training program: 2 sessions of 60 minutes per week, with the focus of the first session on cardiovascular exercises, and the focus of the second session on mobility and strengthening exercises
  Interventions: Other: Exercise program
- control (No Intervention): no intervention (wait and see approach)

INTERVENTIONS:
Other: Exercise program — educational video on training program design and healthy lifestyle 24 training sessions (12 on cardiovascular endurance training, 12 on mobility and strength)
  Arms: Intervention

SUMMARY:
The purpose of this study is to assess the effect of a general training program and educational session to prevent neck and/or low back pain in desktop workers

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all subjects that met the preset inclusion criteria and gave written informed consent to participate will be randomized into an intervention or control group in a 1:1 ratio. Next, subjects of both groups will undergo baseline testing (online survey). The subjects of the intervention group receive a single educational video (online) and are motivated to follow 2 training sessions of 60 minutes each, during 12 consecutive weeks. Instructions for the specific exercises are provided via an online platform. The subjects of the control group are instructed to maintain their normal working activities and activities of daily life and receive no further intervention. Subjects of both groups are prompted to fill out a weekly online logbook to gather information on their physical activity and neck and/or back complaints. All subjects undergo post-intervention testing at 12 weeks (short term effects), 6 months, and 12 months (long term effects).

ELIGIBILITY:
Inclusion Criteria

* age between 18-69 years
* perform regular desktop work (at least 20 hours/week)
* perform desktop work for at least 1 year (employee or student)

Exclusion Criteria:

* documented structural neck- and/or back pathology (confirmed by medical imaging)
* known shoulder or vestibular pathology
* whiplash-associated disorders
* history of surgery in the neck, shoulder, hip, and/or back area
* (history of) chronic pain condition
* serious headache
* serious cardiovascular/metabolic/systemic/neurological conditions
* chronic fatigue syndrome
* fibromyalgia
* psychiatric conditions or history of serious depression
* serious catastrophizing thoughts
* pregnancy or delivery in the past year

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
neck pain | 1 year
  Did you develop neck pain (YES or NO)
low back pain | 1 year
  Did you develop low back pain (YES or NO)

SECONDARY OUTCOMES:
behavioral change | 1 year
  Tendency to remain physically active (PA) during working hours as compared to before your participation in this study (Likert-type scale: not at all PA - slightly less PA - equally PA - slightly more PA - clearly more PA)
physical activity (Baecke Questionnaire) | 1year
  physical activity measurement (activities are scored on a scale of 1-5 with the total scored from 3-15. the lower the score, the less physically active)
time to exposure | 1year
  amount of desktop work (hours/week)
global perceived effect | 1year
  What is your global perceived effect of the intervention program (NRS - score/100)
use of (pain) medication and/or (para)medical care | 1year
  use of (pain) medication and/or (para)medical care (name, dosage/frequency, effect, prescribed or direct acces)
Depression Anxiety Stress Scale-21 (DASS-21 questionnaire) | 1year
  fear, depressive mood, and stress due to COVID-19 crisis and confinement (21 items, Each item is scored from 0 to 3 and is doubled so the global ISI score ranges from 0 to 42)
36-Item Short Form Health Survey (SF-36 questionnaire) | 1year
  quality of life during confinement and telework (item scores are summed to scale scores and transformed into a hundred point scale; scores are transformed so that a higher score indicates better health status)
Insomnia severity index (ISI questionnaire) | 1year
  quality of sleep during confinement and telework (7 items, Each item is scored from 0 to 4 and the global ISI score ranges from 0 to 28)

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No